CLINICAL TRIAL: NCT01854879
Title: Evaluation of Nucleus 6 Sound Coding Algorithms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT004
Record Dates: First submitted 2013-05-13; First posted 2013-05-16 (Estimated); Results first posted 2020-11-04 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Hearing Loss
Keywords: background noise; speech performance; wind noise
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nucleus 6 (Experimental)
  Interventions: Device: Nucleus 6 sound processor

INTERVENTIONS:
Device: Nucleus 6 sound processor

SUMMARY:
The purpose of the study was to evaluate the features of the Nucleus 6 Sound Processor (CP900 series) on existing Nucleus recipients who currently use the previous generation sound processor, the Cochlear Nucleus CP810 (also commonly known as the Nucleus 5), with a Cochlear Nucleus CI24RE, CI512 or CI422 cochlear implant. The features evaluated included an enhanced Automatic Gain Control (eAGC), the option to provide acoustic amplification in combination with traditional electric stimulation through an acoustic component, and three input processing algorithms: Signal to Noise Ratio - Noise Canceller (SNR-NC), Wind Noise Reduction (WNR) and Automatic Scene Analyzer (SCAN).

As is customary for a single-subject research design, study results will be analyzed for each subject individually. For evaluations where testing took place under two conditions (i.e. Endpoint 2, 3, 4, and 5) a non-inferiority hypothesis test based on the paired comparisons of the % of words correct will be performed. For each subject, the paired difference (P1 minus P2) will be calculated and the mean difference will be tested statistically against a non-inferiority null hypothesis of 10%. Successful rejection of the null hypothesis allows for a conclusion that the performance under the test condition 2 (based on the Nucleus 6 sound processor) will be non-inferior to the test condition 1 (based on the Nucleus 5 sound processor).

Ho: P1 - P2 ≥ 10% Ha: P1 - P2 < 10%

We hypothesize acceptance of the null hypothesis for the Nucleus 6 features.

Testing will be based on a paired t-test with a one-sided 0.05 alpha level. The value of 10% was selected as the non-inferiority margin as one that can be tested with reasonable power and was clinically meaningful.

ELIGIBILITY:
Inclusion Criteria:

1. Eight years of age or older
2. CI24RE, CI500 or CI422 series Nucleus cochlear implant types (commercially approved)
3. At least 3 months experience with the cochlear implant
4. Post-linguistic onset of bilateral sensorineural hearing loss, with no congenital component to the hearing loss
5. Native speaker of English, the language used to assess speech perception performance
6. Willingness to participate in and to comply with all requirements of the protocol

Exclusion Criteria:

1. Unrealistic expectations on the part of the subject, regarding the possible benefits, risks, and limitations that are inherent to the prosthetic device 2. Unwillingness or inability of the candidate to comply with all investigational requirements 3. Additional handicaps that would prevent or restrict participation in the audiological evaluations

-

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2013-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Nucleus 6: Nucleus 6 sound processor
Period: Overall Study
Arm/Group | Nucleus 6
Started | 97 (97 consented)
Completed | 92 (92 had matched endpoint data)
Not Completed | 5
Not completed — Could not complete testing within the scheduled time. | 1
Not completed — screen fail | 3
Not completed — incomplete data set | 1

BASELINE CHARACTERISTICS:
Arm/Group | Nucleus 6
Number analyzed (Participants) | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (21.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 49

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Words Correct on AzBio Sentences in Noise S0N90
Description: Individuals were tested with AzBio Sentences in Noise using a speech front (0 degrees) and noise presented to the implant ear (90 degrees) using the following features: enhanced Automatic Gain Control (eAGC), Signal to Noise Ratio - Noise Canceller (SNR-NC), Wind Noise Reduction (WNR) and Automatic Scene Analyzer (SCAN).
Time Frame: Each assessment was completed acutely which equated to approximately 2 hours of testing
Population: subjects enrolled who met candidacy criteria that had paired results for endpoint testing
Measure: Mean (Standard Deviation); unit: percentage of words correct
Arm/Group | Nucleus 6
Number analyzed (Participants) | 92
percentage of words correct | 72.1 (13.6)

ADVERSE EVENTS:
Time Frame: 1 day - study was conducted acutely
Arm/Group | Nucleus 6
Serious Adverse Events (participants affected / at risk) | 0/92
Other Adverse Events (participants affected / at risk) | 0/92

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No